CLINICAL TRIAL: NCT05453370
Title: A Randomized 3-Month, Parallel-Group, Controlled Trial of CALMA M-Health App as an Adjunct to Therapy for the Reduction of Suicidal and Non-Suicidal Self-Injurious Behaviors in Adolescents
Brief Title: CALMA App as an Adjunct to Therapy for Reduction of Suicidal and Non-Suicidal Self-Injurious Behaviors in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Demian Emanuel Rodante, Principal Investigator, University of Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 884
Record Dates: First submitted 2022-06-19; First posted 2022-07-12 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Self-Injurious Behavior
Keywords: Self-Injurious Behavior; Mobile Applications; Dialectical Behavior Therapy; Suicide Prevention
MeSH Terms: conditions — Self-Injurious Behavior; Suicide Prevention | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel group, two-arm randomized controlled trial design, which will employ an intervention condition (CALMA app) and a control condition (Treatment as usual -TAU) with a 3-month follow-up for each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALMA app (Experimental): the arm will receive CALMA app and continue with the usual treatment in a mental health service of a public hospital during the 3 months of the study. In the first interview, the CALMA application will be downloaded to the participant's smartphone. In each follow-up interview (30-days and 60-days), the use of the app will be reinforced.
  Interventions: Device: CALMA m-health app
- Treatment As Usual (TAU) (Other): the arm will not receive the app and will continue with the usual treatment in a mental health service of a public hospital during the 3 months of the study.
  Interventions: Other: Treatment As Usual (TAU)

INTERVENTIONS:
Device: CALMA m-health app — CALMA is an app for smartphones that provides evidence-based tools to prevent suicide. Out of Crisis modality consists of 4 sections: Moments, Agenda, Profile and Tips. The I need help modality uses DBT skills presented in a card format. The Problem-solving Card is the first one showed and helps the user to know if the problem that triggered the crisis can be addressed through a problem-solving strategy. If not, the next step is to use the CALMA thermometer (to identify the intensity of the emotion) and the DBT Skills Cards. They are based fundamentally in two groups of DBT skills, emotional regulation and distress tolerance. If distress worsens or does not diminish the Emergency Card is activated, offering the user the option to make one or several calls to emergency contacts and providing the option to use the geolocation function to show all emergency services near the user's location so that he/she can consult personally. All participants will also receive mental health treatment.
  Arms: CALMA app
Other: Treatment As Usual (TAU) — Participants who do not receive the application will continue the usual mental health treatment (psychotherapeutic and/or psychopharmacological) by their usual treating professionals throughout the duration of the study.
  Arms: Treatment As Usual (TAU)

SUMMARY:
Suicide in the second cause of death in subjects between 15 and 24 years of age. Despite the efficacy of interventions for the management of suicidal crises observed in some clinical trials, a crucial aspect for their effectiveness is accessibility. This leaves little time to intervene during the suicidal process. New platforms to provide evidence-based interventions, universally, economically, and quickly are needed. Smartphones appear to be a good alternative considering the high penetration of these devices locally.

The research group carried out a pilot randomized controlled cluster trial with four weeks of follow-up that provided initial evidence on the safety and acceptability of the app for reducing self-injurious thoughts and behaviors when used as an adjunct to conventional Dialectical Behavioral Therapy (DBT). This study conducted with a group of patients who were already undergoing DBT treatment program, and have shown good acceptability of CALMA as an adjunct to therapy targeting suicidal and non-suicidal self-injury behaviors. Although effectiveness was not the main outcome, results revealed a high probability to decrease suicidal outcomes including ideation, suicidal behaviors, Non-Suicidal Self-Injury (NSSI) and thoughts about NSSI in the group that received CALMA compared to the comparison group.

No specific app for adolescents and young people is available in Spanish. The research group developed CALMA (the Spanish word for "calm"), the first user-interactive mobile app in Spanish. It provides evidence-based tools to manage a suicidal or non-suicidal self-directed violence crisis. CALMA also interacts with the user between crises by promoting activities that reduce their vulnerability to suicide by provide psychoeducation about suicide and its prevention. Based on these encouraging initial findings, in this project the investigators propose to scale the intervention to a larger group of patients, focus it on adolescents and including public hospitals not specialized in DBT.

This is a parallel group, two-arm randomized controlled trial design, which will employ an intervention condition (CALMA app) and a control condition (Treatment as usual) with a 3-month follow-up for each participant, to evaluate the effectiveness, safety and acceptability of CALMA, a suicide prevention app for smartphones, to reduce the frequency of self-injurious thoughts and behaviors in adolescents who are assisted in a Mental Health service of three Public Hospitals.

DETAILED DESCRIPTION:
Suicide and suicidal behaviors are among the leading causes of death and injury worldwide. Although in Argentina the overall suicide rate has remained relatively stable in the last 15 years, when analyzing the rates by age group, it is observed that in that same period there was a gradual and sustained growth in the suicide rate in subjects between 15 and 24 years of age. Despite the efficacy of interventions for the management of suicidal crises observed in some clinical trials, a crucial aspect for their effectiveness in daily practice is accessibility, that is, the availability of the intervention at the time of the crisis. This leaves little time to intervene during the suicidal process. This is why, beyond employing effective interventions to prevent suicide, it is necessary that they be quickly accessible at the time of crisis. New platforms to provide evidence-based interventions, universally, economically, and quickly are needed. Smartphones appear to be a good alternative considering the high penetration of these devices locally. The development of mobile applications (apps) for the prevention of suicidal behavior is recent.

The research group carried out a pilot randomized controlled cluster trial with four weeks of follow-up that provided initial evidence on the safety and acceptability of the app for reducing self-injurious thoughts and behaviors when used as an adjunct to conventional Dialectical Behavioral Therapy (DBT). This study conducted with a group of patients who were already undergoing DBT treatment program, have shown good acceptability of CALMA as an adjunct to therapy targeting suicidal and non-suicidal self-injury behaviors. Furthermore, although effectiveness was not the main outcome, results revealed a high probability to decrease suicidal outcomes including ideation, suicidal behaviors, Non-Suicidal Self-Injury (NSSI) and thoughts about NSSI in the group that received CALMA compared to the comparison group To investigators knowledge, no specific app for adolescents and young people is available in Spanish. The research group developed CALMA (the Spanish word for "calm"), the first user-interactive mobile app in Spanish. CALMA provides evidence-based tools to manage a suicidal or non-suicidal self-directed violence crisis with the goal of preventing death by suicide. CALMA also interacts with the user between crises by promoting activities that reduce their vulnerability to suicide by provide psychoeducation about suicide and its prevention. Based on these encouraging initial findings, in this project the investigators propose to scale the intervention to a larger group of patients, focus it on adolescents and include public hospitals not specialized in DBT.

The investigators are conducting a parallel group, two-arm randomized controlled trial design, which will employ an intervention condition (CALMA app) and a control condition (Treatment as usual -TAU) with a 3-month follow-up for each participant, to evaluate the effectiveness, safety and acceptability of CALMA, a suicide prevention app for smartphones, to reduce the frequency of self-injurious thoughts and behaviors in adolescents who are assisted in a Mental Health service of three Public Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 10 to 19 years old who come on an outpatient basis or have been hospitalized in Mental Health Services
* Have a smartphone where the application can be installed and used are eligible to participate in the study
* Have attempted suicide, or exhibited a suicidal gesture or self-injurious behavior (according to the SITBI definition) in the last month before entering the study
* Agree to give their informed consent and their guardian agrees to sign your informed consent

Exclusion Criteria:

* If the participant plans not to continue the treatment in the next 3 months or
* Has an inability to provide assent/consent for cognitive or language reasons
* Do not have the functional capacity to use the application, which will be operationally determined by a score below 30 on the Self-Care motor domain, below 10 on the Communication cognitive domain or below 14 on the Cognitive domain of Social Knowledge in the Functional Independence Measurement scale (FIM).

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency of Suicidal and Non-Suicidal Self-Injurious Behaviors. | Participants will be assessed at four timepoints: day-0 (baseline), day-30, day-60 and day-90.
  Suicidal behavior will be assessed using the Spanish version of the Self-Injurious Thoughts and Behaviors Interview (SITBI). This is a structured interview consisting of 169 items divided into 5 modules that examine the presence, frequency and characteristics of 5 types of self-injurious behavior: a) suicidal ideation; b) suicide plans; c) suicidal gestures; d) suicide attempts and e) self-harm. The SITBI conceptualizes suicide risk on a continuum, starting with suicide ideation (SI) ("thoughts of killing yourself?"), possibly accompanied by a suicide plan ("think about how you might kill yourself [e.g., taking pills, shooting yourself] or work out a plan of how to kill yourself?") and in some cases by suicide attempt (SA) ("made a suicide attempt [i.e., purposefully hurt yourself with at least some intent to die]?"). The construction of the questions in the original SITBI are consistent with the commonly accepted definitions of each type of behavior.

SECONDARY OUTCOMES:
Levels of Emotional Dysregulation | Participants will be assessed at two timepoints: day-0 (baseline) and day-90.
  Emotional dysregulation will be quantified with the Spanish version of the Emotional Regulation Difficulties Scale (DERS). It has 36 items with a Likert-type response format (from 1 = almost never to 5 = almost always) and a six-factor structure: 1) Impulse control difficulties; 2) Limited access to emotional regulation strategies; 3) Non-acceptance of emotional responses; 4) Difficulty engaging in goal-directed behavior; 5) Lack of emotional awareness; 6) Lack of emotional clarity. The DERS has previously been used in pre- and post-intervention studies as an emotional dysregulation state variable to assess effectiveness. This variable has eleven reverse-scored items and will be considered as a quantitative variable (minimum value = 80; maximum value = 136). Higher scores suggest greater problems with emotion regulation.
Levels of Engagement of the app. | Participants will be assessed at three timepoints: day-30, day-60, and day-90.
  The use of the app will be obtained and recorded via an objective measure recorded from the participant's phone number. Specifically, use will be considered when at least one of the following features of CALMA is used during the study period: opened a "Tips", arrived at the "Emergency Card", finished a crisis (due to success or abandonment), opened a notification, added a contact, reviewed their "Moments", added a picture or content to their "Moments", closed the app while it was in crisis and ended a crisis successfully. Patients will be defined as "users" of the app if they met the following criteria: subjectively reported using the app in the survey and used at least one feature recorded by our objective measures.

OTHER OUTCOMES:
Time (days) to psychiatric admission | from the date of enrollment to the date of the first psychiatric hospitalization for a self-injurious behavior up to 3 months. Participants will be assessed at the three follow-up timepoints: day-30, day-60, and day-90.
  At follow-ups and at the final interview, participants will be asked if they have had a psychiatric hospitalization for a self-injurious behavior during the follow-up period. This measure will be used to compare time to psychiatric admission in those participants who received the intervention with those participants who did not receive the app.
Sociodemographic variables | Participants will be assessed at day-0 (baseline).
  Sociodemographic variables are: age, sex, gender, sexual orientation, education level and treatment modality (outpatient/inpatient).

CONTACTS AND LOCATIONS:
Overall Officials: Demián E Rodante, MD, MsC, Principal Investigator — Institute of Pharmacology, School of Medicine, University of Buenos Aires; Federico M Daray, MD, MsC, PhD, Study Director — Institute of Pharmacology, School of Medicine, University of Buenos Aires
Locations (4):
- Argentina (4):
  - Pedro de Elizalde Children's General Hospital, City of Buenos Aires, Buenos Aires
  - Institute of Pharmacology of the School of Medicine of the University of Buenos Aires, City of Buenos Aires, Buenos Aires
  - Interzonal Acute Hospital "San Roque" de Gonnet, La Plata, Buenos Aires
  - Children's Hospital "Sor María Ludovica", La Plata, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daray FM, Olivera Fedi RH, Rodante DE. [Development of CALMA: A mobile APP for the prevention of suicide in adolescents and youth]. Vertex. 2018 Jan;29(137):55-64. Spanish. PMID 30605196
- [Background] Rodante DE, Kaplan MI, Olivera Fedi R, Gagliesi P, Pascali A, Jose Quintero PS, Compte EJ, Perez AI, Weinstein M, Chiapella LC, Daray FM. CALMA, a Mobile Health Application, as an Accessory to Therapy for Reduction of Suicidal and Non-Suicidal Self-Injured Behaviors: A Pilot Cluster Randomized Controlled Trial. Arch Suicide Res. 2022 Apr-Jun;26(2):801-818. doi: 10.1080/13811118.2020.1834476. Epub 2020 Oct 18. PMID 33073745
- [Derived] Rodante DE, Chiapella LC, Olivera Fedi R, Papavero EB, Lavoie KL, Daray FM. A randomized 3-month, parallel-group, controlled trial of CALMA m-health app as an adjunct to therapy to reduce suicidal and non-suicidal self-injurious behaviors in adolescents: study protocol. Front Psychiatry. 2023 Jul 20;14:1087097. doi: 10.3389/fpsyt.2023.1087097. eCollection 2023. PMID 37547219
- See also: Official educational and non-profit web page of the CALMA app where the functioning of the app is described. — https://www.appcalma.com/